CLINICAL TRIAL: NCT01465074
Title: Effects of Acute Nicotine on Long-term Potentiation in the Dorsolateral Prefrontal Cortex of Patients With Schizophrenia and Healthy Controls
Brief Title: Effects of Acute Nicotine Treatment on Neuroplasticity and Memory in Patients With Schizophrenia
Acronym: NIC-PAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited staff and operating resources
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tony George, Professor, MD, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NICPAS#024/2011
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Schizophrenia
Keywords: nicotine; memory; plasticity; TMS; Paired Associative Stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine gum (4 mg) (Active Comparator): Nicotine gum will be given once on one of the two test days in a randomized, double-blinded fashion. Gum will be chewed for 30 min before the plasticity induction occurs.
  Interventions: Drug: Nicotine polacrilex
- Regular Mint Gum (Placebo Comparator): Regular, taste-, texture- and color matched with the Nicotine Gum will be ingested once on one of the two testing days, 30 min before plasticity induction.
  Interventions: Drug: Regular chewing gum; Dentyne Ice, Wrigely´s Mint Gum

INTERVENTIONS:
Drug: Nicotine polacrilex — 4 mg
  Other Names: Nicorette, Extreme Chill
  Arms: Nicotine gum (4 mg)
Drug: Regular chewing gum; Dentyne Ice, Wrigely´s Mint Gum — 30 min chewing, one dose
  Arms: Regular Mint Gum

SUMMARY:
Patients with schizophrenia display cognitive impairments, such as reduced attention and problems with memory. Available medications for schizophrenia poorly alleviate memory problems however, research indicates that nicotine improves memory. In order for there to be memories formed, there has to be changes (neuroplasticity changes) in how the brain cells communicate. One way to induce such changes is by using Transcranial Magnetic Stimulation (TMS) combined with peripheral nerve stimulation in a Paired Associative Stimulation (PAS) paradigm. The investigators laboratory has developed a novel method that measures memory-like brain changes using electroencephalography (EEG), TMS and PAS. The present study will use this novel method to evaluate the effects of acute nicotine gum (4mg) and placebo (regular) gum on memory and memory-like brain changes in schizophrenia and healthy controls. The hypothesis is that nicotine will improve memory and facilitate neuroplasticity changes in the prefrontal cortex of patients with schizophrenia to a larger extent than in healthy controls.

DETAILED DESCRIPTION:
Background: Schizophrenia (SCZ) is frequently associated with marked working memory (WM) deficits whose pathophysiology is closely related to dorsolateral prefrontal cortex (DLPFC)-dependent dysfunction[1]. These deficits predict disease outcome and poor response to antipsychotic treatment[2]. Consequently, elucidating the physiology of DLPFC-dependent WM deficits in SCZ is key in better understanding this illness and its treatment.

Patients with SCZ display an unusually high prevalence of smoking and high rates of smoking cessation failures are commonly associated with WM deficits[3]. The central nicotinic acetylcholine receptor (nAChR) is the main target for nicotine. Several lines of evidence strongly suggest that the nAChR system is a promising target for treating cognitive deficits in SCZ. These include the following observations: (1) expression of nAChRs receptors is abnormal in several brain regions, including the PFC, in post mortem brains of patients with SCZ, (2) genes coding for nAChR subunits are candidate risk genes for SCZ and nicotine addiction, and (3) smoking abstinence produce deficits of WM, which correlate with blood levels of nicotine, are alleviated by smoking re-instatement and are blocked by nAChR antagonists in patients with SCZ, but not in healthy control smokers (e.g.,[4]). However, the underlying mechanism through which nicotine and nAChRs affect DLPFC-dependent memory in SCZ are still unknown. Nicotine-induced increases in neural plasticity may represent one such mechanism.

Neuroplasticity, which includes long-term potentiation (LTP), is a proposed physiological mechanism for memory formation. LTP is dependent on an optimal interaction between the glutamate (GLU), dopamine (DA) and γ-Aminobutyric acid (GABA) systems and perturbations in these systems likely explain why patients with SCZ demonstrate deficits in WM and neuroplasticity[5,6]. nAChR are present on GABA, GLU and DA neurons and nicotine could potentially improve cognition by modulating these systems. Studies have demonstrated that acute nicotine administration potentiates neural plasticity in the motor cortex of healthy human subjects. One of these studies used Paired Associative Stimulation (PAS), a powerful paradigm to index LTP in the motor cortex, to assess the effects of nicotine on LTP in non-smokers[7]. The results demonstrate that nicotine enhanced LTP-like mechanisms induced by PAS in the motor cortex[7]. To date, however, there has been no direct measure of LTP-like plasticity from the DLPFC in humans. To overcome this challenge, the investigators group has developed a novel PAS technique of combined transcranial magnetic stimulation (TMS) and electroencephalography (EEG)[8] to directly index LTP from the DLPFC.

Conventional methods of applying PAS involves the repetitive delivery of two paired stimulations: the first being an electrical peripheral nerve stimulation of the right median nerve of the hand and 25 ms later a second TMS pulse delivered to the contralateral motor cortex (hence PAS-25). Through repetitive pairing of these two stimulations, PAS-25 results in increased activation of output neurons that represents a direct measure LTP in humans[9]. The investigators lab has recently recorded PAS-LTP in the DLFPC using a novel technique of TMS-EEG[8]. Here, PAS is applied to the DLPFC by repetitive delivery of: (1) a peripheral nerve stimulation to the right side, followed 25 ms later by; (2) a TMS pulse delivered to the left DLPFC. PAS-induced potentiation of cortical evoked activity is then measured directly from the DLPFC and represents LTP in this region as interneurons activated from cortical stimulation and peripheral stimulation, in turn, activate DLPFC output neurons contemporaneously and increase their activity when repeated over 30 min. Thus, the activation of the somatosensory cortex by peripheral nerve stimulation will propagate to the DLPFC and arrive there simultaneously with the TMS pulse resulting in LTP. The validity of this technique relies on the observation that there are strong correlations between TMS induced evoked potentials in the motor and DLPFC (r=0.8-0.85, p<0.001)[8]. LTP is quantified as change in DLPFC cortical evoked activity from baseline (pre-PAS) to different time points following PAS-25 (post-PAS). Preliminary data from the investigators ongoing study using these novel methods, demonstrate that PAS-25 induces significant LTP in the DLPFC. For example, in healthy controls cortical evoked activity in the DLPFC was facilitated by 56% post-PAS (maximal point of facilitation) while in patients with SCZ the cortical evoked activity post-PAS was only increased by 16% (Cohen's d=0.80). This is to the investigators knowledge the first time LTP has ever been demonstrated in-vivo in the DLPFC of humans and the first time that LTP deficits in the DLPFC have been reported in patients with SCZ. The aim of this proposal is now to assess whether enhanced WM by nicotine is mediated by potentiation of LTP in the DLPFC.

Hypothesis:

1. Patients with SCZ will have reduced DLPFC LTP and impaired WM compared to healthy controls.
2. Acute nicotine gum challenge will attenuate the DLPFC LTP and WM deficit in patients with SCZ.
3. Plasma nicotine levels will correlate with improvement in DLPFC LTP.
4. Reversal of the DLPFC LTP deficit in patients with SCZ will be associated with improvement in WM.

Methods:

Subjects: Fourteen healthy non-smokers and 14 non-smokers with SCZ will complete this exploratory study. This sample size is based on a previous study that used the TMS-EEG method and demonstrated a significant difference in cortical inhibition between healthy controls and SCZ patients[10], and will be sufficient to detect a medium effect size (Cohen´s d=0.72; α=0.05, 1-β=0.80) of nicotine treatment. Only patients that are treated with a stable dose of antipsychotic medication (≥1 month) will be enrolled in this study. This could potentially confound the results as the investigators are using healthy non-medicated controls for comparison. However, the within- subjects design is an effort to control for such effects. Study design: The study will be a double-blinded, placebo-controlled, crossover study consisting of two PAS-25 testing sessions one month apart, followed by a 7 day post-PAS follow-up test session each. Pharmacological treatment: Nicotine (4 mg) or matching placebo gum will be administered on each of the two test days before baseline TMS-EEG recording. Maximum nicotine blood concentration is reached after 30 min, at which point blood samples will be drawn to assess nicotine levels. WM assessment: The N-back task measures the ability to maintain active information online (i.e. WM) and is dependent on DLPFC functioning. Letters are presented in a continuous sequence and the subject is asked to respond if they recognize the present letter as the same letter appears that appeared as the N (0, 1, 2 or 3) letters back, i.e. "N-back". The N-back will be administered at the pre-test training session (to control for training effects), baseline, 120 minutes and 1 week post PAS. Paired Associative Stimulation (PAS): The pairings will occur over a 30 min period and the peripheral nerve stimulation and TMS to the DLPFC will be delivered at 0.1 Hz. To assure the DLPFC localization, neuronavigational techniques using the MRIcro/reg software and a T1-weight MRI scan will be used. Quantifying LTP: To assess DLPFC LTP, change in cortical evoked activity will be measured using pre- and post-PAS TMS-EEG recordings. TMS pulses will be generated using two Magstim 200 stimulators (Magstim Company Ltd., UK) connected to and a 7 cm figure-of-eight coil via a Bistim module. A train of 100 pulses (0.1 Hz) will be administered together with EEG recordings; (1) before PAS in order to assess baseline cortical evoked activity and (2) at different time points (0, 15, 30, 60,120 min and 7 days) following PAS-25. EEG will be recorded using the DLPFC-corresponding electrodes of a 64-channel Synamps 2 EEG system. Cortical evoked activity will be defined as the area under the rectified curve for the averaged EEG recordings (50-275 ms post-stimulus) and LTP will be quantified as the change in cortical evoked activity from baseline. Statistics: Within and between subjects comparisons will be carried out using repeated measures, mixed-factorial, ANOVAs when appropriate. Relationship between LTP and nicotine levels will be assessed using Pearson correlations. P-values will be set to 0.05 and multiple comparisons will be Bonferroni corrected.

Significance: The results of this study will provide important new knowledge about mechanisms underlying cognitive enhancement strategies in SCZ. That is, the investigators intend to decipher the complex pharmacological mechanisms that underlie nicotinic cholinergic enhancement of plasticity in the DLPFC. Such findings will also help to generate important biomarkers through which cognitive enhancing strategies may be measured biologically that can potentially lead to the development of more personalized treatments of cognitive deficits in this debilitating disorder.

ELIGIBILITY:
Inclusion criteria:

* Age of 18-55 years
* Non-smoker or past smoker, abstinent for at least the last 1 year, non-smoking status will be assessed on the test days by saliva cotinine levels <15ng/mL and exhalation CO levels <10ppm.
* Females with potential childbearing must have a negative urine pregnancy test at inclusion.
* Women with child-bearing potential must use contraceptives during the trial Acceptable means of contraception are hormonal methods (pill, injection, vaginal ring), male or female condom, abstinence, injectable contraceptives, intrauterine devices or abstinence.
* Ability and willingness to speak English
* Willingness to provide informed consent
* Adequate hearing and visual capacity, or corrected by visual/ hearing aid • Right handedness

Patients with schizophrenia:

* Current diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV TR criteria
* Stable antipsychotic treatment or dosage for the past 4 weeks prior to study entry
* Clinically stable, i.e. no psychotic episode that required hospitalization within the last 3 months prior to study inclusion

Exclusion Criteria:

General

* Current smoker or abstinent smoker for less than 1 year
* Past or current history of drug abuse disorder or current elicit drug use, positive urine drug screen (for any other drug besides benzodiazepines) on any of the two test days
* Current or past history of neurological disorder, i.e. meets criteria for a cognitive disorder secondary to a neurological or other medical disorder affecting the central nervous system (such as, traumatic brain injury, stroke, Parkinson).
* Current or past history of seizures
* Any metal implants
* Mini Mental Status Examination score of ≤17
* Diagnosis of bipolar disorder or current major depressive episode
* Electroconvulsive Therapy (ECT) within 6 months prior to study participation
* Allergy to any of the following: nicotine resin, xylitol, butylhydroxythyolen E 321, sodium carbonate, corn starch, magnesium oxide, D&C Yellow No 10, menthol, acesulfam potassium, wax, titan oxide, maltitol, sorbitol, gum base, sucralose, palm oil, mannitol, glycerin, calcium carbonate, gum arabic.
* Any of the following; breast feeding, immediate post-myocardial infarction period, life-threatening arrhythmias, angina pectoris, and active temporomandibular joint disease, oral or pharyngeal inflammation, or history of esophagitis or peptic ulcer.

Healthy controls:

* Any psychiatric diagnosis except for simple phobias or an adjustment disorder as diagnosed by DSM IV TR
* Psychotropic medication (except for sedative /hypnotics at a stable dose for at least 4 weeks).
* Sedative /hypnotics at a stable dose less than 4 weeks
* A first-degree relative with as past or present history of primary psychotic disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in prefrontocortical neuroplasticity | 0, 15, 30, 60, 120 min, 7 days post treatment
  Change in cortical evoked activity (using EEG) from baseline to the different time points following paired associative stimulation.

SECONDARY OUTCOMES:
Change in working memory | baseline, 30 and 120 min and 7 days post treatment
  N-back performance can be assessed in four conditions, where 0-back is the control condition in which the test subject responds to every letter that appears on the screen, making sure the person can respond to the stimuli as it requires no on-line retention of information. The 1, 2 and 3 back conditions assess on-line retention with increasing difficulty. Average performance, i.e. number of accurate responses as well as response time, will be used as outcome measures.
  PAS-NBACK=(Average performance Post-PAS/ Average performance at baseline)*100

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, M.D., Principal Investigator — Centre for Addiction and Mental Health, Schizophrenia Program, Toronto, ON, Canada; Jeff Z Daskalakis, M.D., Ph.D., Principal Investigator — Centre for Addiction and Mental Health, Brain Stimulation Lab, Toronto, ON, Canada
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Weinberger DR, Berman KF, Zec RF. Physiologic dysfunction of dorsolateral prefrontal cortex in schizophrenia. I. Regional cerebral blood flow evidence. Arch Gen Psychiatry. 1986 Feb;43(2):114-24. doi: 10.1001/archpsyc.1986.01800020020004. PMID 3947207
- [Background] Green MF. Cognitive impairment and functional outcome in schizophrenia and bipolar disorder. J Clin Psychiatry. 2006;67 Suppl 9:3-8; discussion 36-42. PMID 16965182
- [Background] Moss TG, Sacco KA, Allen TM, Weinberger AH, Vessicchio JC, George TP. Prefrontal cognitive dysfunction is associated with tobacco dependence treatment failure in smokers with schizophrenia. Drug Alcohol Depend. 2009 Sep 1;104(1-2):94-9. doi: 10.1016/j.drugalcdep.2009.04.005. Epub 2009 May 17. PMID 19447570
- [Background] Wing VC, Sacco KA, George TP. Spatial working memory impairments induced by cigarette smoking abstinence are correlated with plasma nicotine levels in schizophrenia. Schizophr Res. 2011 May;128(1-3):171-2. doi: 10.1016/j.schres.2010.10.011. Epub 2010 Nov 13. No abstract available. PMID 21075601
- [Background] Lewis DA, Gonzalez-Burgos G. Neuroplasticity of neocortical circuits in schizophrenia. Neuropsychopharmacology. 2008 Jan;33(1):141-65. doi: 10.1038/sj.npp.1301563. Epub 2007 Sep 5. PMID 17805309
- [Background] Daskalakis ZJ, Christensen BK, Fitzgerald PB, Chen R. Dysfunctional neural plasticity in patients with schizophrenia. Arch Gen Psychiatry. 2008 Apr;65(4):378-85. doi: 10.1001/archpsyc.65.4.378. PMID 18391126
- [Background] Thirugnanasambandam N, Grundey J, Adam K, Drees A, Skwirba AC, Lang N, Paulus W, Nitsche MA. Nicotinergic impact on focal and non-focal neuroplasticity induced by non-invasive brain stimulation in non-smoking humans. Neuropsychopharmacology. 2011 Mar;36(4):879-86. doi: 10.1038/npp.2010.227. Epub 2010 Dec 15. PMID 21160466
- [Background] Farzan F, Barr MS, Levinson AJ, Chen R, Wong W, Fitzgerald PB, Daskalakis ZJ. Reliability of long-interval cortical inhibition in healthy human subjects: a TMS-EEG study. J Neurophysiol. 2010 Sep;104(3):1339-46. doi: 10.1152/jn.00279.2010. Epub 2010 Jun 23. PMID 20573972
- [Background] Stefan K, Kunesch E, Cohen LG, Benecke R, Classen J. Induction of plasticity in the human motor cortex by paired associative stimulation. Brain. 2000 Mar;123 Pt 3:572-84. doi: 10.1093/brain/123.3.572. PMID 10686179
- [Background] Farzan F, Barr MS, Levinson AJ, Chen R, Wong W, Fitzgerald PB, Daskalakis ZJ. Evidence for gamma inhibition deficits in the dorsolateral prefrontal cortex of patients with schizophrenia. Brain. 2010 May;133(Pt 5):1505-14. doi: 10.1093/brain/awq046. Epub 2010 Mar 28. PMID 20350936
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research